CLINICAL TRIAL: NCT06043583
Title: Intrauterine Device Versus Uterine Artery Embolization for Adenomyosis: A Randomized Controlled Trial Comparing Therapeutic Efficacy
Brief Title: Intrauterine Device Versus Uterine Artery Embolization for Adenomyosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0729
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Intrauterine Devices; Uterine Artery Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrauterine device (Active Comparator)
  Interventions: Procedure: Intrauterine device
- Uterine artery embolization (Active Comparator)
  Interventions: Procedure: Uterine artery embolization

INTERVENTIONS:
Procedure: Intrauterine device — The vagina is visually inspected to check the size and position of the uterus. The speculum is inserted into the vagina. The IUD is placed inside the uterus and then the strings are cut.
  Arms: Intrauterine device
Procedure: Uterine artery embolization — The right common femoral artery is punctured under ultrasound guidance and a 5F vascular sheath is inserted into the Rt common femoral artery. A 5F catheter was inserted into the internal iliac artery, and a 2.0F microcatheter is advanced into the uterine artery. Embolization is performed using polyvinyl alcohol (PVA). One third (20 mL) of a 60-mL mixture comprising 150-250-µm PVA particles was injected at the beginning of embolization into each uterine artery, followed by injection of at least two thirds (40 mL) to all (60 mL) of a mixture comprising 250-355- µm PVA particles and finally completion with 355-500- µm PVA particles. Embolization was performed until complete cessation of blood flow in the ascending uterine artery for 10 heart beats.
  Arms: Uterine artery embolization

SUMMARY:
The primary purpose of this study is to compare the therapeutic efficacy of intrauterine device and uterine artery embolization for uterine adenomyosis.

DETAILED DESCRIPTION:
Screening

* History, Physical examination
* Laboratory test (Hemoglobin) / MRI
* Pictorial blood loss assessment chart
* Symptom/Quality of life score

Intervention

* Intrauterine device or uterine artery embolization
* Adverse event montoring

Follow-up visit #1 (1 month)

* Vital signs
* blood test (Hemoglobin) / Ultrasound
* Adverse event monitoring

Follow-up visit #2 (3 month)

• MRI only for embolization patients

Follow-up visit #3 (6 months)

* Blood test (Hemoglobin) / Ultrasound
* Pictorial blood loss assessment chart
* Symptom/Quality of life score

Follow-up visit #4 (12months)

* Blood test (Hemoglobin) / Ultrasound
* Pictorial blood loss assessment chart
* Symptom/Quality of life score

ELIGIBILITY:
Inclusion Criteria:

1. Women with symptomatic fibroids (age: 19 - 48 years old) 2. Hemglobin < 12g/dL, 3. Symptoms of adenomysis (Menorrhagia, Dysmenorrhea)

Exclusion Criteria:

1. Gynecologic malignancy 2. Ongoing infection or inflammation 3. Coagulopathy (platelet < 50,000 or INR > 1.5) 4. Concomitant endometriosis 5. Pregnancy

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | Hemoglobin level at 6 and 12 months after each procedure
  Hemoglobin as an indicator of menstrual bleeding

SECONDARY OUTCOMES:
Pictorial blood loss assessment chart (PBAC) | 0,6,12 months
  Pictorial blood loss assessment chart: a semi-quantitative method for evaluation of menstrual blood loss (>100 considered as heavy mentrual blood)
Visual analogue scale | 0,6,12 months
  Visual analogue scale: a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
Symptom and quality of life score questionnaire | 0,6,12 months
  Symptom and quality of life score questionnaire: a questionnaire developed to objectively assess symptom severity and quality of life in relation to uterine adenomyosis before and after procedure
Uterine volume | 0,12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No